CLINICAL TRIAL: NCT01043809
Title: Evaluation of a School-based Handwashing Promotion Program in Three Countries
Brief Title: Evaluation of a Handwashing Promotion Program in Three Countries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Procter and Gamble (Industry); Zhejiang Provincial Center for Disease Control and Prevention (Other Government); Centers for Disease Control and Prevention, China (Other Government); Project HOPE (Unknown); Field Epidemiology Training Program Alumni Foundation, Inc. (Other)
Responsible Party: Anna Bowen, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCEZID-5281
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Infectious Disease; Respiratory Illness; Absenteeism
Keywords: schools; handwashing; prevention and control; communicable diseases; absenteeism
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Randomly selected schools will not receive handwashing intervention
- 2 (Experimental): Randomly selected schools will get standard commercial school-based handwashing promotion
  Interventions: Behavioral: Procter & Gamble school-based handwashing promotion program
- 3 (Experimental): Randomly selected schools will receive standard commercial school-based handwashing promotion program, plus an added level of handwashing promotion (varies by country)
  Interventions: Behavioral: expanded school-based handwashing promotion

INTERVENTIONS:
Behavioral: Procter & Gamble school-based handwashing promotion program — Handwashing promotion lesson and materials targeting first grade students
  Arms: 2
Behavioral: expanded school-based handwashing promotion — Procter & Gamble's standard school-based handwashing promotion education and materials targeting first grade students, plus a program enhancement. In China, enhancement consists of a supply of soap for school sinks. In Pakistan, enhancement consists of soap for school sinks, plus enlistment of a peer hygiene champion in each first grade class. In the Philippines, enhancement consists of enlistment of a peer hygiene champion in each first grade class.
  Arms: 3

SUMMARY:
The purpose of this study is to assess whether simple, school-based handwashing promotion impacts health and hygiene knowledge among students and their families.

ELIGIBILITY:
Inclusion Criteria:

* 19 students per first grade class

  * Piped water tap available to every 30 first grade students for handwashing

Exclusion Criteria:

* Compulsory handwashing or distribution of hand wipes before school lunch
* Commercial handwashing promotion at school during previous 5 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
student school absences / 100 student-weeks of observation | one semester

SECONDARY OUTCOMES:
Student absences due to respiratory illness / 100 student-weeks of observation | one semester
student absences due to infectious syndromes / 100 student-weeks of observation | one semester
longitudinal prevalence of infectious syndromes among students' family members | one semester

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bowen, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (3):
- Zhejiang Province CDC, Hangzhou, Zhejiang, China
- Project HOPE, Karachi, Sindh, Pakistan
- FETPAFI, Manila, Philippines